CLINICAL TRIAL: NCT00618683
Title: Localization of the Anterograde and Retrograde Components of the Reentrant Circuit of AV Nodal Reentrant Tachycardia
Brief Title: AV Nodal Reentrant Tachycardia Study
Acronym: AVNRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2353; AHA (Other: American Heart Association)
Record Dates: First submitted 2008-02-07; First posted 2008-02-20 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Tachycardia, Atrioventricular Nodal Reentry
Keywords: AVNRT; Atrioventricular; nodal reentrant circuit; nodal reentrant tachycardia; Paroxysmal supraventricular tachycardia
MeSH Terms: conditions — Tachycardia, Atrioventricular Nodal Reentry; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Arm (Other): Mapping and Ablation
  Interventions: Procedure: Cardiac Invasive Electrophysiological Study

INTERVENTIONS:
Procedure: Cardiac Invasive Electrophysiological Study — Mapping and localizing of the components of the reentrant circuit as part of the Electrophysiological Study

SUMMARY:
The purpose of this study is to determine/identify what mechanisms/factors are involved with regard to AV nodal reentrant tachycardia.

DETAILED DESCRIPTION:
HYPOTHESES:

1. The Tendon of Todaro forms a line of block during slow/fast AVNRT preventing the atrial impulse from entering the triangle of Koch (and perhaps providing sufficient time for activation to pass through the coronary sinus coat to activate the posterior extensions of the AV node as is critical to maintenance of tachycardia)
2. The coronary sinus myocardial coat participates in all of the forms of AVNRT. The reentrant circuit is thus not confined within the triangle of Koch and sites remote from the compact AV node could be targeted for ablation reducing the risk of AV conduction block.
3. A model of the reentrant circuit can be created for each patient's tachycardia, using the site of earliest retrograde activation to suggest the retrograde limb and the resetting response to suggest the anterograde limb.

DATA ANALYSIS/STATISTICS:

Resetting and Mapping of AV nodal reentrant tachycardia:

Pacing will be analyzed to see at which sites, the tachycardia can be reset by the latest extra-stimuli (i.e., with the least advancement in local activation). The coupling interval will be compared to the latest extra-stimulus capable of resetting (advancing) the tachycardia from the postero-septal tricuspid annulus.

Ablation Results:

The patients will act as their own reference, since the standard ablation technique in the postero-septal space is being performed first and tested for efficacy. The McNemar test will be applied to compare the efficacy of ablation at the postero-septal tricuspid annulus alone (standard ablation), with the efficacy of this ablation plus ablation within the coronary sinus. From our initial observations, It is anticipated that the additional ablation in the coronary sinus will increase the efficacy of the procedure from <95% to >98%, such that 100 cases should provide sufficient data to reach statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-80
* At least one documented episode of AV nodal reentrant tachycardia
* Patient scheduled for electrophysiology study and catheter ablation for supraventricular tachycardia

Exclusion Criteria:

* Ages < 16 or > 80
* Medical condition significantly increasing risk of extending procedure time or X-ray exposure
* Pregnancy
* Prior ablation with radiation exposure >2 hours
* Electrophysiology study performed without sedation or anesthesia
* Unavailable for follow-up

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2004-03-25 (Actual); Primary Completion 2020-01-21 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
raise the frequency of success to more than 98% | unk

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavrakis, MD, Principal Investigator — University of Oklahoma
Locations (1):
- The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States